CLINICAL TRIAL: NCT00146289
Title: A Randomised, DB, Placebo-controlled, Parallel Group, 16-wk MICARDIS (160mg) Tab, Proof-of-concept, Evaluating Insulin Sensitivity in Overweight or Obese, Non-diabetic, Normotensive, Using the OGTT, With a Clamp Sub-group
Brief Title: The Primary Objective of This Study is to Determine Whether MICARDIS® Improves Insulin Sensitivity in Overweight or Obese, Non-diabetic, Normotensive Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.469
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Telmisartan

INTERVENTIONS:
Drug: MICARDIS® (telmisartan)

SUMMARY:
The primary objective of this study is to determine whether MICARDIS® improves insulin sensitivity in overweight or obese, non-diabetic, normotensive subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation.
2. Subjects 18-65 years old.
3. Body Mass Index (BMI) >= 28.
4. Sedentary life style defined as: Does not engage in vigorous activity for more than 30 minutes per day, more than two times per week.
5. Waist circumference >= 40 inches (102 cm) in men and >= 35 inches (89 cm) women.
6. HbA1C assessed <= 6.5%.
7. Triglycerides >= 150, and <= 500 mg/dL.
8. Fasting Glucose <= 126 mg/dL.
9. Blood pressure >= 110/64 and <= 140/90 mmHg.

Exclusion Criteria:

1. Currently taking any antihypertensive medications (e.g., thiazide or loop diuretics), diabetic medications, medications known to alter insulin sensitivity (e.g., statins), steroids, glucocorticoids, niacin, nicotinic acid, and anti-psychotic/depressant drugs (e.g., prozocin). Including over the counter (OTC) and herbal products, which are known to affect metabolic function.
2. Diagnosis of any of the following chronic diseases: hypertension, diabetes mellitus, renal insufficiency, congestive heart failure, hepatic insufficiency, biliary obstructive disorders, autoimmune disease, HIV, coronary artery disease, mental illness, and severe anemia.
3. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator.
4. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve.
5. Unstable angina or myocardial infarction or cardiac surgery within the past 3 months.
6. PCI (percutaneous coronary intervention) within the past 3 months.
7. Stroke within the past 6 months.
8. Bilateral renal artery stenosis or obstructive disorders, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney.
9. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT (ALT) or SGOT (AST) > 2.5 times the upper limit of normal range, or
   * Serum creatinine > 2.3 mg/dL (or > 203 mol/L)
10. Pre-menopausal women (last menstruation <=1 year prior to signing informed consent) who:

    * Have a positive urine pregnancy test (UPT) prior to randomisation (Visit 2 or Visit 2.1 for subject participating in the clamp procedure)
    * Are not surgically sterile, or
    * Are nursing, or pregnant, or
    * Are of child-bearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the study and do not agree to periodic pregnancy testing during participation in the study. Acceptable methods of birth control are limited to: Intra-Uterine Device (IUD), oral, implantable or injectable contraceptives and estrogen patch. No exceptions will be made.
11. Hematocrit < 35%.
12. Primary aldosteronism.
13. Hereditary fructose intolerance.
14. History of drug or alcohol dependency within the previous 6 months.
15. Currently participating in a weight loss program.
16. Any investigational drug therapy within one month of randomisation or during the study.
17. Known hypersensitivity to any component of the study drug (telmisartan or placebo).
18. Any circumstances the Investigator feels participation in the study would hinder subject safety or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138
Dates: Start 2005-02; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline to the end of study (16 weeks) in the insulin sensitivity index as estimated by the composite index (R04-1184) calculated from a 3-hour oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
From baseline: Glucose disposal rates; Insulin sensitivity (IS) index as Rd/I (clamp); IS index (OGTT- min model); Insulin secretion capacity; fasting insulin & gluc.; AUC gluc & insulin; ratio of AUC glucose ÷ by AUC insulin; lipids & inflam. markers.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (17):
- United States (8):
  - UCLA School of Medicine- Divison of Endocrinology, Los Angeles, California
  - University of CA at SanDiego- Department of Endocrinology, San Diego, California
  - Boehringer Ingelheim Investigational Site, Westlake Village, California
  - Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - University of Rochester Medical Center, Rochester, New York
  - Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - Boehringer Ingelheim Investigational Site, Harker Heights, Texas
- Canada (3):
  - University of Manitoba, Diabetes Research Group, Winnipeg, Manitoba
  - St. Joseph's Health Care London, London, Ontario
  - The Ottawa Hospital - Riverside Campus, Ottawa, Ontario
- Århus Sygehus, Aarhus C, Denmark
- Germany (3):
  - Universitätsmedizin Berlin, Berlin
  - Boehringer Ingelheim Investigational Site, Künzing
  - Boehringer Ingelheim Investigational Site, Unterschneidheim
- Italy (2):
  - Policlinico Monteluce, Perugia
  - Azienda Ospedale Università di Pisa, Pisa